CLINICAL TRIAL: NCT05734534
Title: Effects of BFR Interventions on Muscle Function and Adaptations in Healthy Individuals and Individuals With COPD
Brief Title: Effects of BFR Interventions in Healthy Individuals and Individuals With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BFR
Record Dates: First submitted 2022-12-23; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy; COPD
Keywords: BFR; COPD; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BFR-ST and BFR-HIT (Experimental): Participants will be allocated to a BFR intervention including resistance training and high-intensity intervals performed on a bicycle ergometer, both performed with BFR.
  Interventions: Other: BFR during training
- HL-ST and HIT (Active Comparator): Participants will be allocated to heavy load resistance training and high-intensity intervals performed on a bicycle ergometer, both performed without BFR
  Interventions: Other: BFR during training
- BFR-P (Experimental): Participants with COPD experiencing an acute exacerbation of their COPD requiring hospitalization will be allocated to application of BFR twice daily throughout their hospitalization. Participants are resting in a supine position throughout the application of BFR.
  Interventions: Other: BFR during rest
- BFR-NMES (Experimental): Participants with COPD experiencing an acute exacerbation of their COPD requiring hospitalization will be allocated to application of BFR with neuromuscular electrical stimulation (BFR-NMES) twice daily throughout their hospitalization. Participants are resting in a supine position throughout the application of BFR-NMES.
  Interventions: Other: BFR during rest
- Control group (Active Comparator): Participants with COPD experiencing an acute exacerbation of their COPD requiring hospitalization will allocated to usual care, consisting of daily physiotherapy sessions.
  Interventions: Other: BFR during rest

INTERVENTIONS:
Other: BFR during training — Healthy participants and participants diagnosed with COPD will be randomized to either the BFR-ST and BFR-HIT or to HL-ST and HIT
  Arms: BFR-ST and BFR-HIT; HL-ST and HIT
Other: BFR during rest — Participants experiencing acute exacerbation of their COPD requiring hospitalization will be randomized to either BFR-P, BFR-NMES or the control group throughout their hospitalization.
  Arms: BFR-NMES; BFR-P; Control group

SUMMARY:
The purpose of the study is to investigate the effect of different blood flow restriction (BFR) interventions on muscle function and adaptations both in healthy well-trained individuals and individuals diagnosed with COPD.

ELIGIBILITY:
Inclusion criteria for participants with COPD group are:

* Diagnosis with COPD

Exclusion criteria participants in the COPD group are

* Having experienced an acute exacerbation of COPD within the last 6 weeks (Study A)
* Taking part in pulmonary rehabilitation within the last 3 months (Study A)
* Presenting with a history of thromboembolic event in the lower limbs.

Inclusion criteria for healthy participants are:

* Age between 18 and 40 years.
* Maximal oxygen uptake (VO2max) of >55 ml O2/kg/min for men and >50 ml O2/kg/min for women
* BMI of <26 and normal ECG and blood pressure.

Exclusion criteria for healthy participants are:

* Smoking
* chronic disease,
* Use of prescription medication
* Pain due to current or previous musculoskeletal injury
* Resistance training more than once per week in the 12 months leading up to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Change assessed from before to after the intervention (6 weeks in study A, on average 7 days in study B)
  Maximal voluntary isometric contraction of m. quadriceps femoris

SECONDARY OUTCOMES:
Lean mass | Change assessed from before to after the 6 week intervention
  Lean mass assessed by dual X-ray absorptiometry (DXA)
Maximal oxygen consumption | Change assessed from before to after the 6 week intervention
  VO2max during incremental exercise
Skeletal muscle mitochondrial respiration | Change assessed from before to after the intervention (6 weeks in study A, on average 7 days in study B)
  High resolution respirometry
Fiber cross-sectional area | Change assessed from before to after the intervention (6 weeks in study A, on average 7 days in study B)
  Immunohistochemistry to determine fiber cross-sectional area
Myonuclei | Change assessed from before to after the intervention (6 weeks in study A, on average 7 days in study B)
  Immunohistochemistry to determine number of myonuclei
Functional exercise capacity | Change assessed from before to after the 6 week intervention (only in individuals with COPD)
  Number of repetitions achieved during a 1-minute sit-to-stand test
Satellite cells | Change assessed from before to after the intervention (6 weeks in study A, on average 7 days in study B)
  Immunohistochemistry to determine number of satellite cells

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided